CLINICAL TRIAL: NCT01779297
Title: New Integrated Weaning Indexes From Mechanical Ventilation: A Prospective Clinical Trial
Brief Title: New Integrated Weaning Indexes
Acronym: NIWIs
Status: Completed | Type: Observational
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Senior Intensivist Nurse, Phd Candidate in Nursing, Baqiyatallah Medical Sciences University
Other Study IDs: BMSU & TUMS
Record Dates: First submitted 2013-01-23; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Mechanical Ventilation Weaning
Keywords: new integrative weaning indexes; mechanical ventilation; ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether introducing the new weaning indexes can predict better than traditional ones?

DETAILED DESCRIPTION:
The study was divided into two parts: First, the threshold values of the indexes that discriminated best between successful weaning and weaning failure were determined in training set (n = 208). Second, the accuracy of each index was scrutinized prospectively in an additional group of patients (prospective-validation data set, n = 967). One thousand one hundred and seventy-five patients who were on mechanical ventilation for more than 24 hours were evaluated.Informed consent was obtained from each patient, whenever possible, or from the patient's next of kin. The samples were selected using a simple random sampling method in which the entry number of eligible patients was considered to be the sampling ID number. Using Random Allocation Software (RAS), random numbers were generated to select the study participant.

The ventilators used were Evita XL and Evita 4 edition (Draeger, Lubeck, Germany).

According to a protocol that have introduced in two studies, the protocol established. All of the mechanically ventilated patients undergoing assessment for extubation undergo a daily SBT if predetermined eligibility criteria for weaning are met . According to this protocol, sedation would be discontinued before evaluation of weaning. Patients who meet these criteria are initially placed on SBT (continuous positive airway pressure of 5 mmHg, FiO2≤0.4) for 3 minutes to obtain weaning parameters. If the Oxygen saturation is ≥ 92% on pulse oximetry with FiO2≤0.4 and RSBI <104 breaths/minute/L, patients are continued on the SBT for 30 to 120 minutes. All clinical and ventilator parameters are monitored closely for signs of respiratory distress (respiratory rate > 30 breaths/minute, SaO2< 90%, heart rate > 140 breaths/minute, or a sustained increase or decrease of heart rate of >20%, blood pressure>200 mm Hg or <80 mm Hg, and agitation, diaphoresis, or anxiety). At the end of the SBT, the RSBI is measured again, ABG is obtained, and the predetermined values are calculated and measured. The decision to return to mechanical ventilation made by the two subspecialists in pulmonary and lung diseases, who were chief supervisor of both ICU in two cities (who were completely blind to the study and the results of the indexes evaluated), based on airway competence (cough, sputum production, neurologic status, level of consciousness, and maximal inspiratory pressure). Patients who remain extubated at 48 hours are classified as having had a successful extubation. Baseline demographics, initial diagnosis, and pre-extubation clinical, ventilator, laboratory, and radiographic data are collected for each patient.

To assess the prognostic value of new indices, receiver operator characteristic (ROC) curves was drawn for each formula in addition for other conventional criteria used in this area. For each ROC curve analysis, sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value, diagnostic accuracy, likelihood ratio of a positive test (LR+) and the likelihood ratio of a negative test (LR-), probability for weaning success when test is positive and probability for weaning success when test is negative of the indexes were used to predict the weaning outcome in the prospective-validation data set.

Hanley and McNeil method was used to calculate the area under curve (AUC) for each formula and then the methods developed by the same authors were used to compare these AUCs. Bayes' theorem was used to compute the weaning outcome the probability for weaning success when test is positive and negative (post-test probability) in the prospective-validation data set to assess the perform

ELIGIBILITY:
Inclusion Criteria:

* Patients (both males and females) more than 24 hours in mechanical ventilation in weaning process.

Exclusion Criteria:

1. Hypercapnic respiratory failure attributable to COPD exacerbation or post-respiratory arrest;
2. underlying moderate to severe obstructive airways disease, defined as forced expiratory volume in 1 second of < 50% of predicted value, or baseline PaCO2 > 50 mmHg,
3. concurrent neurological and neuromuscular or drug intoxication contributing to respiratory failure; and finally younger than 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One thousand one hundred and seventy-five patients who were on mechanical ventilation for more than 24 hours were evaluated.
Sampling Method: Probability Sample
Enrollment: 1175 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Better accuracy in predicting weaning outcome | Four years

SECONDARY OUTCOMES:
Adequate prognosis | Four years
  The following measurements were taken for weaning indexes:
  1. RSBI
  2. NIF
  3. P0.1
  4. CROP
  5. IWI
  6. PaO2: PALVO2 ration (PPR)
  7. PaO2:FiO2 ratio (PFR)
  8. RR
  9. VT
  10. MV
  11. C Dynamic
  12. C Static
  13. Pimax
  14. PaO2
  15. PaCO2
  16. FiO2
  17. SaO2
  18. Respiratory index
  19. Formula one [(PPR)/ (RSBI*FiO2)]
  20. Formula two [(PPR)/ (RSBI*FiO2*P0.1)]
  21. Formula three [(PPR)*(NIF)/ (RSBI*FiO2)]
  22. Formula four [(PPR)*(NIF)/ (RSBI*FiO2*P0.1)]
  23. Formula five [(NIF)/ (P0.1)]
  24. Formula six [(SaO2)/ ((P (A-a) O2)*RSBI*FiO2)]
  25. Formula seven [(SaO2)/ ((P (A-a) O2)*RSBI*FiO2*P0.1)]
  26. Formula eight [(SaO2*NIF)/ ((P (A-a) O2)*RSBI*FiO2)]
  27. Formula nine [(SaO2*NIF)/ ((P (A-a) O2)*RSBI*FiO2*P0.1)]
  28. Formula ten [(SaO2)/ ((P (A-a) O2)*P0.1)] These are newly proposed indexes, used in some hospitals in Iran.

CONTACTS AND LOCATIONS:
Locations (1):
- Shariati hospital, Mousavi Hospital, Valiasr hospital, Tehran & Zanjan, Iran